CLINICAL TRIAL: NCT06931912
Title: Growth Evaluation, Health Promotion, and Clinical Management in Children and Adolescents With Thalassemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMSCRF2024041
Record Dates: First submitted 2025-01-07; First posted 2025-04-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-04

CONDITIONS: Thalassemia Intermedia; Thalassemia Major; Growth Delay; Puberty, Delayed
Keywords: Thalassemia; Children and adolescents; Growth development; Health Promotion; Clinical Management
MeSH Terms: conditions — beta-Thalassemia; Puberty, Delayed; Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric patients with growth problems (Experimental): We identify pediatric patients with growth problems by conducting growth and development assessments. Implement the MENBS clinical interventions for pediatric patients with growth problems.
  Interventions: Behavioral: MENBS clinical interventions

INTERVENTIONS:
Behavioral: MENBS clinical interventions — * Monitor: Continuously monitor health-related indicators through regular follow-up.
  * Education: Provide health education to improve cognition of patients and their families.
  * Nutrition: Assess patients' nutritional risks and develop personalized diet plans.
  * Behavior: Recommend appropriate exercise plans to promote physical development.
  * Support: Conduct home visits, offer free clinics and establish a support network.

SUMMARY:
There are nearly 300,000 patients with severe or intermediate thalassemia in China. Growth retardation is the most significant health issue for children and adolescents with transfusion-dependent thalassemia (TDT), placing a substantial economic burden on their families and a serious social strain on the labor force. Investigating the growth and development of these children and adolescents, and establishing targeted intervention plans, holds significant social value for public health practice.

1. To screen and identify pediatric patients with growth problems by conducting growth and development assessments in high-incidence areas of China, including physical development, endocrine function, nutritional status, brain function and lifestyle behaviors.
2. Implement the MENBS clinical interventions for pediatric patients with growth problems, concentrating on the following areas:

   * Monitor: Continuously monitor health-related indicators through regular follow-up.
   * Education: Provide health education to improve the cognition of patients and their families.
   * Nutrition: Assess patients' nutritional risks and develop personalized diet plans.
   * Behavior: Recommend appropriate exercise plans to promote physical development.
   * Support: Conduct home visits, offer free clinics and establish a support network.
3. Repeat growth assessment for pediatric patients with growth problems after 1-year clinical interventions.
4. Evaluate the effectiveness of MENBS interventions by comparing changes in growth and development indicators.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with transfusion-dependent thalassemia (TDT)
* Male or female age ≤18 years
* Subjects who are willing and able to provide written informed consent

Exclusion Criteria:

* Not applicable

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 369 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Height-for-age (m) | Up to 1 year
  It is assessed using the 'Growth Standard for Children under 7 Years of Age' and the 'Standard for Height Level Classification among Children and Adolescents Aged 7-18 Years' issued by the National Health Commission
Body mass index-for-age (BMI-for-age, kg/m^2) | Up to 1 year
  It is assessed using the 'Growth Standard for Children under 7 Years of Age' and the 'Dietary Guidelines for Chinese Residents'.
Puberty status | Up to 1 year
  Puberty status will be measured using by Tanner scale (TS). It is a five-stage system to assess breast development (in girls), genital development (in boys), pubic hair growth (in both sexes).
Endocrine function | Up to 1 year
  Endocrine function such as hormonal levels (IGF-1, GH, etc.) will be measured by clinical examination
Nutritional status | Up to 1 year
  Nutritional status will be measured by clinical examination, such as concentration of Vitamin D and Zinc
Intelligence quotient (IQ) | Up to 1 year
  IQ will be measured by scores obtained from Raven's Progressive Matrices. Raw scores are converted into percentile ranks or IQ scores based on age-group norms:
  * ≥95th percentile (IQ ~125+): Very high intelligence.
  * 75th-94th percentile (IQ ~110-124): Above average.
  * 25th-74th percentile (IQ ~90-109): Average range (most common).
  * 5th-24th percentile (IQ ~80-89): Below average.
  * <5th percentile (IQ <80): Potential intellectual disability.
Brain function | Up to 1 year
  Brain function will be measured by Functional Near-infrared Spectroscopy (fNIRS) to record brain activations
Quality of life | Up to 1 year
  Quality of life will be measured using by Pediatric Quality of Life Inventory (PedsQL), with higher scores indicating better quality of life. The score range is 0-100.

CONTACTS AND LOCATIONS:
Locations (1):
- Regenerative Medicine Center and Red Blood Cell Disorders Center, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No